CLINICAL TRIAL: NCT02548806
Title: Randomised Single Dose 3 Way Crossover Single Blind Study to Evaluate the Pharmacokinetic Dose Proportionality, Compare the Bioavailability and Safety of Clonidine Mucoadhesive Buccal Tablets (MBT) With Catapres in Normal Healthy Volunteers
Brief Title: Phase 1 PK, Bioavailability, Safety Study of Clonidine MBT w Catapres in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OX2015/28/02
Record Dates: First submitted 2015-09-02; First posted 2015-09-14 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Clonidine
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clonidine MBT 50µg (Experimental): Each subject will receive the following treatments in random order over 3 Treatment Periods (1 treatment/period): Clonidine MBT 50µg single dose, Clonidine MBT 100μg single dose ,a single-dose of reference catapres 100μg tablets.
  Interventions: Drug: Clonidine MBT 50µg
- Clonidine MBT 100µg (Experimental): Each subject will receive the following treatments in random order over 3 Treatment Periods (1 treatment/period): Clonidine MBT 50μg single dose, Clonidine MBT 100µg single dose ,a single-dose of reference catapres 100μg tablets..
  Interventions: Drug: Clonidine MBT 100µg
- Catapres 100μg (Active Comparator): Each subject will receive the following treatments in random order over 3 Treatment Periods (1 treatment/period): Clonidine MBT 50μg single dose, Clonidine MBT 100μg single dose ,a single-dose of reference catapres 100μg tablets.
  Interventions: Drug: Catapres 100μg

INTERVENTIONS:
Drug: Clonidine MBT 50µg — Clonidine MBT 50µg, single dose
  Other Names: Clonidine Lauriad
  Arms: Clonidine MBT 50µg
Drug: Clonidine MBT 100µg — Clonidine MBT 100µg, single dose
  Other Names: Clonidine Lauriad
  Arms: Clonidine MBT 100µg
Drug: Catapres 100μg — Catapres tablet 100μg, single dose
  Other Names: Catapres
  Arms: Catapres 100μg

SUMMARY:
The purpose of this study is to determine the pharmacokinetic dose proportionality of 50 μg and 100 μg Clonidine and comparative bioavailability of clonidine with that from the Reference drug, Catapres® 100 μg oral tablets following single dose administration in healthy subjects.

DETAILED DESCRIPTION:
A single blind, randomised, 3-period, 3-sequence single-dose crossover study to determine the pharmacokinetic dose proportionality of Clonidine MBT 50 μg and Clonidine MBT 100 μg and comparative bioavailability of clonidine from the Reference drug, Catapres® 100 μg oral tablets following single dose administration in healthy male and female subjects.

36 subjects will be randomised for 30 to complete the study. The study will comprise of 3 Treatment Periods (1, 2 and 3) and a post study follow up (7 - 12 days after the last dose). Study drug will be administered on the morning of Day 1. Pharmacokinetic (PK) blood samples will be collected for each of three treatment periods. Safety will be evaluated at specified times throughout the study. There will be at least 7 days between dose administrations.

ELIGIBILITY:
Main Inclusion Criteria:

* Healthy males or females (non-pregnant/non-lactating) aged 18 - 50 years.
* A Body Mass Index (BMI) of 18-30.
* No clinically significant abnormal serum biochemistry, haematology and urine examination values.
* A negative urinary drugs of abuse screen.
* Negative HIV and Hepatitis B and C results.
* No clinically significant abnormalities in 12-lead electrocardiogram (ECG).
* No clinically significant abnormalities in blood pressure or pulse.
* No allergy or sensitivity to clonidine or any of its excipients.
* No allergy to milk or milk derivatives.
* Subjects must provide written informed consent to participate in the study

Main Exclusion Criteria:

* Current or past medical condition that might significantly affect the pharmacokinetic or
* pharmacodynamic response to clonidine.
* Participation in a New Chemical Entity clinical study within the previous 3 months or a marketed drug clinical study within the previous 30 days.
* Pathological condition of the oral cavity that would affect administration via the buccal route.
* Raynaud's disease or other peripheral vascular disease.
* Receipt of regular medication within 14 days of the first dose that may have an impact on the safety and objectives of the study (at the Investigator's discretion).
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
* Symptomatic postural hypotension evident on screening
* History or evidence of Suicidal Ideation and/or behaviour as determined by using Columbia-Suicide Severity Rating Scale (C-SSRS)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Dose proportionality of two strengths of clonidine MBT (50μg and 100 μg) as assessed by Non-compartmental pharmacokinetic analysis (Area Under the Curve) | 3 Months
  To evaluate dose proportionality of two strengths (50 μg and 100 μg) of Clonidine MBT, by using Area Under the Curve (AUC)
Bioavailability of clonidine from Clonidine MBT 50 μg and 100 μg with that from oral clonidine hydrochloride 100 μg tablets. (Area Under the Curve) | 3 Months
  To compare the bioavailability of clonidine from Clonidine MBT® 50 μg and 100 μg with that from oral clonidine hydrochloride 100 μg tablets, by using Area Under the Curve (AUC)

SECONDARY OUTCOMES:
General safety information (adverse events, (AEs), 12-lead electrocardiogram (ECG) and vital signs), during the study period. | 3 Months
  Number of Participants With Treatment-Related Adverse Events as Assessed by Common Toxicity Criteria for Adverse Effects (CTCAE v4.0), 12-lead electrocardiogram (ECG) and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, MD, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Limited, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
presentation at ESMO congress

REFERENCES:
- [Derived] Vasseur B, Dufour A, Houdas L, Goodwin H, Harries K, Emul NY, Hutchings S. Comparison of the Systemic and Local Pharmacokinetics of Clonidine Mucoadhesive Buccal Tablets with Reference Clonidine Oral Tablets in Healthy Volunteers: An Open-Label Randomised Cross-Over Trial. Adv Ther. 2017 Aug;34(8):2022-2032. doi: 10.1007/s12325-017-0585-9. Epub 2017 Jul 19. PMID 28726169